CLINICAL TRIAL: NCT01236638
Title: A Phase II, Open-Label Extension Study Evaluating the Long Term Safety, Tolerability & Efficacy of Orally-Administered CYT387 in Primary Myelofibrosis or Post-Polycythemia Vera or Post-Essential Thrombocythemia Myelofibrosis
Brief Title: Extension Study Evaluating the Long Term Safety and Efficacy Study of CYT387 in Primary Myelofibrosis (PMF) or Post-polycythemia Vera (PV) or Post-essential Thrombocythemia (ET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCL09101E
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis
Keywords: Primary Myelofibrosis; Post-Polycythemia Vera; Post-Essential Thrombocythemia; CYT387 (momelotinib)
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Momelotinib (Experimental)
  Interventions: Drug: Momelotinib

INTERVENTIONS:
Drug: Momelotinib — Patients will continue receiving the same doses as assigned during the CCL09101 protocol; up to 400 mg once per day (QD). CYT387 will be administered orally as a single daily dose (at least 20 and no more than 28 hours apart, preferably in a fasted state at least two hours before and one hour after a meal), except for patients on the twice daily (BID) dosing regime (150 mg BID).
  Other Names: CYT387

SUMMARY:
This extension protocol to the core study CCL09101 allows patients who have tolerated the drug and derived a clinical benefit, to continue to receive treatment beyond the 9 cycles of the core protocol. Long term safety and efficacy of CYT387 (momelotinib) will be evaluated.

DETAILED DESCRIPTION:
The myeloproliferative neoplasms (MPN), most notably polycythemia vera (PV), essential thrombocythemia (ET), and primary myelofibrosis (PMF) are a diverse but inter-related suite of clonal disorders of pluripotent hematopoietic stem cells (Tefferi et al., 2008). The MPN share a range of biological, pathological, and clinical features including the relative overproduction of one or more cells of myeloid origin, growth factor independent colony formation in vitro, marrow hypercellularity, extramedullary hematopoiesis, spleno- and hepatomegaly, and thrombotic and/or hemorrhagic diatheses (Tefferi et al., 2005).

This is a multi centre, open-label, extension study of the core study (CCL09101). The primary aims of the study will be to determine the long term safety and tolerability of orally-administered CYT387 when administered as a capsule dose, on a 28-day treatment cycle.

Following completion of the core study (CCL09101), patients who have tolerated the drug and derived clinical benefit will continue to be treated with CYT387 administered orally.

Subjects will be evaluated every three months for up to 24 cycles of CYT387 treatment. Subjects will return for a follow-up visit 30 days after completion of the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed at least 9 cycles of treatment on the core study 'A Phase I/II, Open-Label, Dose-Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally-Administered CYT387 in Primary Myelofibrosis or Post-Polycythemia Vera or Post-Essential Thrombocythemia Myelofibrosis (CCL09101)' and achieved stable disease (SD), clinical improvement (CI), partial remission (PR) or complete remission (CR) using the International Working Group consensus criteria for treatment responses in myelofibrosis with myeloid metaplasia (IWG-MRT; Tefferi et al., 2006)
* Must be able to provide informed consent and be willing to sign an informed consent form.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Must have evidence of acceptable organ function within 7 days of initiating study drug as evidenced by the following:

  * SGOT (AST) or SGPT (ALT) <= 2.5 x upper limit of normal (ULN) (or <= 5 x ULN if in the investigator's opinion the elevation is due to extramedullary hematopoiesis)
  * Bilirubin <= 2.0 x ULN or direct bilirubin < 1.0
  * Serum creatinine <= 2.5 x ULN
  * Absolute neutrophil count >= 500/µL
  * Platelet count >= to 20,000/µL
* Females of childbearing potential must have a negative pregnancy test within 4 days of entering the extension protocol.

Exclusion Criteria:

* A delay of 4 weeks or more since the last preceding dose of CYT387 on the CCL09101 core study.
* Any chemotherapy (e.g., hydroxyurea), immunomodulatory drug therapy (e.g., thalidomide), immunosuppressive therapy, corticosteroids > 10 mg/day prednisone or equivalent, or growth factor treatment (e.g., erythropoietin) within 14 days prior to initiation of study drug.
* Incomplete recovery from major surgery within four weeks of study entry.
* Radiation therapy within four weeks of study entry.
* Women of childbearing potential, unless surgically sterile for at least 3 months (i.e., hysterectomy), OR postmenopausal for at least 12 months (FSH > 30 U/mL), OR unless they agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through end of study. Permitted methods for preventing pregnancy must be communicated to study subjects and their understanding confirmed.
* Men who partner with a woman of childbearing potential, unless they agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through to the end of study. Permitted methods for preventing pregnancy must be communicated to study subjects and their understanding confirmed.
* Females who are pregnant or are currently breastfeeding.
* Known positive status for HIV.
* Clinically active hepatitis B or C.
* Diagnosis of another malignancy unless free of disease for at least three years following therapy with curative intent. Patients with early-stage basal cell or squamous cell skin cancer, cervical intraepithelial neoplasia, cervical carcinoma in situ or superficial bladder cancer may be eligible to participate at the Investigator's discretion.
* Any acute active infection.
* Cardiac dysrhythmias requiring treatment, or prolongation of the QTc (Fridericia) interval to >450 msec for males or >470 msec for females at pre-study screening, unless attributable to pre-existing bundle branch block.
* Presence of >= Grade 2 peripheral neuropathy.
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), uncontrolled or unstable angina, myocardial infarction, cerebrovascular accident, or pulmonary embolism within 3 months prior to initiation of study drug.
* Uncontrolled inter current illness or any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine the long term safety and tolerability of orally-administered CYT387 in patients with PMF or post-ET/PV MF following completion of core study CCL09101 | Safety monitoring will be undertaken for all patients every 3 months
To obtain information on the long term effectiveness of orally-administered CYT387 in patients with PMF or post-ET/PV MF | Every three months
  Measured by complete response (CR) rate, partial response (PR) rate and clinical improvement (CI) rate according to IWG-MRT consensus criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ayalew Tefferi, MD, Study Chair — Mayo Clinic
Locations (6):
- United States (3):
  - Stanford Cancer Center, Stanford, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
- The Royal Melbourne Hospital, Parkville, Victoria, Australia
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec